CLINICAL TRIAL: NCT06909409
Title: D Vitamin and Alveolar Macrophages in Idiopathic Pulmonal Fibrosis
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 1-10-72-166-23
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-10

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
Keywords: Idiopathic pulmonary fibrosis; pulmonary macrophages; alveolar macrophages; vitamin D; Soluble CD163; Soluble CD206
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood: Serum and EDTA-plasma. Bronchoalveolar lavage fluid (BALf). Cryobiopsy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with IPF
- Patients with non-IPF interstitial lung disease (ILD)
- Patients with lung cancer

SUMMARY:
The goal of this observational study is to gain deeper insights into human macrophages and vitamin D, and their interplay, within Idiopathic Pulmonary Fibrosis (IPF).

The overall questions, it aims to answer, are the following:

Do IPF patients suffer from systemic and local (pulmonary) insufficient levels of vitamin D? Do IPF patients suffer from pro-fibrotic and pro-inflammatory pulmonary macrophages?

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of IPF, non-IPF ILD or lung cancer
* A signed informed consent

Exclusion Criteria:

* Do not speak Danish/Do not understand Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients at the Department of Respiratory Diseases and Allergy, Aarhus University Hospital, Denmark, diagnosed with ILD or lung cancer.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2026-10-11 (Estimated); Study Completion 2026-10-11 (Estimated)

PRIMARY OUTCOMES:
Vitamin D status | At enrollment
  Significant change in vitamin D levels in systemic (blood) and local (pulmonary) metabolism.
Pulmonary macrophages | At enrollment
  Significant change in alveolar macrophage phenotype

SECONDARY OUTCOMES:
Biomarker levels in blood and BAL samples | At enrollment
  Significant change in levels of macrophage and inflammatory/fibrotic biomarkers

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Denmark, Aarhus N, Denmark